CLINICAL TRIAL: NCT03980093
Title: A Novel Values-Based Intervention to Increase Endocrine Therapy Adherence Among Breast Cancer Survivors
Brief Title: The REACH Study: A Novel Values-Based Intervention to Increase Endocrine Therapy Adherence Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joanna Arch, Associate Professor, Department of Psychology and Neuroscience, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18-0234; R21CA218723 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-06-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education plus Values (Experimental)
  Interventions: Behavioral: Education; Behavioral: Values
- Education (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Online medical education on the benefits of anti-hormonal medication, potential side effects, and how to manage them.
Behavioral: Values — An Acceptance and Commitment Therapy (ACT)-based intervention consisting of brief online sessions plus a visual cue-based intervention focused on personal values.
  Arms: Education plus Values

SUMMARY:
This pilot trial compares two online interventions to improve adherence to anti-hormonal medication among women with the most common form of breast cancer (estrogen receptor-positive).

ELIGIBILITY:
Inclusion Criteria include:

1. Women in Colorado treated for Stage 0 to III estrogen receptor-positive breast cancer who have completed primary cancer treatment (surgery, chemotherapy, and/or radiation) and within the past 2.5 years, have been prescribed anti-hormonal therapy
2. Take their anti-hormonal therapy medication at least occasionally and have at least 1 more year left on their prescription
3. Report at least 1 factor that makes taking their anti-hormonal therapy medication difficult
4. Have internet access

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence assessed by electronic pillbox (Wisepill box) | Change from baseline through 6 month follow-up

SECONDARY OUTCOMES:
Self-reported medication adherence | Change from baseline to 3 and 6 month follow-up
  Reported anti-hormonal medication pills missed, past 30 days, with a validated self-reported medication adherence item
Positive and negative emotional associations with taking anti-hormonal medication | Change from baseline through 6 month follow-up
  Emotional Attitudes Scale, adapted to focus on anti-hormonal medication
Intentions to adhere to anti-hormonal medication in the next year and next several years | Change from baseline through 6 month follow up
  Anti-Hormonal Medication Intentions Scale (average score on a 1 to 7 scale; higher=better outcome, e.g., stronger intentions to adhere), adapted from the Health Behavior Intentions Scale
Medication nonpersistence assessed by electronic pillbox (Wisepill box) | Baseline through 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joanna J Arch, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Rocky Mountain Cancer Centers, Greenwood Village, Colorado, United States